CLINICAL TRIAL: NCT06350500
Title: Addressing Disparities in Breast Cancer Care: An Approach to Health Equity
Brief Title: A Patient Navigation Program for Addressing Disparities in Breast Cancer Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: I-3858823
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Breast Carcinoma; Breast Ductal Carcinoma in Situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Patient Navigation; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Services Research (Patient Navigation) (Experimental): Patients receive patient navigation services from a patient navigator as needed to improve knowledge about clinical and supportive care services, navigate to existing services, help manage barriers to care, and enhance skills related to management of cancer treatment
  Interventions: Behavioral: Patient Navigation; Other: Questionnaire

INTERVENTIONS:
Behavioral: Patient Navigation — Receive patient navigation
Other: Questionnaire — Ancillary studies

SUMMARY:
This clinical trial evaluates a patient navigation program for addressing disparities in breast cancer care. The navigation program is designed to help improve patient knowledge about clinical and supportive care services, navigate to existing services, help manage barriers to care, and enhance patient skills related to management of cancer treatment. Offering a patient navigation program may increase health equity and improve social needs and quality of life over time for newly diagnosed breast cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Implement a patient navigation program in the Roswell Park Breast Clinic focused on underserved women with a first cancer diagnosis of breast cancer or ductal carcinoma in situ (DCIS) (n=126).

SECONDARY OBJECTIVE:

I. Systematically address barriers to care by connecting women with multiple barriers of care with a first diagnosis of breast cancer or DCIS to supportive services and culturally appropriate resources.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Have a confirmed diagnosis of breast cancer or Ductal Carcinoma In Situ (DCIS)
* Currently identify their gender as woman or female
* Was assigned female sex at birth (AFAB)

  - Participant is experiencing ≥1 barrier to care as determined by the social needs screening tool
* Participant must understand the investigational nature of this study and verbally consent to participate prior to receiving any study related intervention

Exclusion Criteria:

* Participants who are not suspected of or diagnosed with breast cancer or Ductal Carcinoma in Situ (DCIS)
* Participants who have had a previous diagnosis of any cancer
* Participants who were assigned male sex or intersex at birth
* Unwilling or unable to follow protocol requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Enrollment rate | Up to 2 years
  Enrollment rate Will be defined as the number of patients enrolled divided by the number of patients approached. The enrollment rate will be estimated with a 90% credible region obtained by Jeffrey's prior method.
Reasons for refusal | Up to 2 years
  Reported reasons of refusal will be summarized using frequencies and relative frequencies
Retention Rate | Up to 2 years
  The number of patients that complete patient navigation divided by the number of patients enrolled
Reasons for discontinuation | Up to 2 years
  Will be summarized using frequencies and relative frequencies

SECONDARY OUTCOMES:
European Organization for Research and Treatment of Cancer Quality of Life Scale (EORTC QLQ-C30) | Up to 2 years
  the quality of life in breast cancer patients. Score averaged, transformed to 0-100 scale, higher score indicates better quality of life
Social Determinates of health | Up to 2 years
  An 11 question survey . A score of 11 or more when the numerical values for answers to questions 7-10 are added shows that the person might not be safe.
Barriers to care | Up to 2 years
  Patient navigators will meet with participants to discuss barriers to care. Results will be summarized
Use of supportive services | Up to 2 years
  Will be summarized using frequencies and relative frequencies
Patient Satisfaction survey | up to 2 years
  Will be summarized (by time as appropriate) using frequencies and relative frequencies

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Glaser, Principal Investigator — Roswell Park Comprehensive Cancer Center
Locations (1):
- Roswell Park Comprehensive Cancer Center, Buffalo, New York, United States